CLINICAL TRIAL: NCT00422214
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, Phase III Study of the Efficacy and Safety of Quetiapine Fumarate (Seroquel SR®) Sustained-Release as Monotherapy in Adult Patients With Acute Bipolar Depression
Brief Title: Phase III/Seroquel SR Bipolar Depression Monotherapy - US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D144CC00002
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Affective Psychosis, Bipolar; Depression, Bipolar; Manic-Depressive Psychosis; Psychoses, Manic-Depressive
Keywords: Bipolar Disorder; Bipolar Depression,; Manic Depression; Seroquel; Seroquel SR; quetiapine fumarate
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate (Seroquel) SR

SUMMARY:
The purpose of this study is to determine the safety and efficacy of sustained-release quetiapine fumarate (Seroquel®) in the treatment of patients with Acute Bipolar Depression for 8 weeks.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Documented diagnosis of Bipolar 1 disorder or Bipolar 11 disorder
* Outpatient status at enrollment

Exclusion Criteria:

* Patients with >8 mood episodes during the past 12 years
* Use of prohibited medications
* Substance or alcohol abuse or dependence
* Current suicide risk or suicide attempt within last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depression symptoms by final visit as measured by the MADRS total score

SECONDARY OUTCOMES:
Change from baseline to final visit on the MADRS total score MADRS item scores, CGI-BP-S, CGI-BP-C

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Datto, MD, Study Director — AstraZeneca; Larisa Acevedo, Ph.D, Study Director — AstraZeneca
Locations (54):
- United States (54):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Cerritos, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Oceanside, California
  - Research Site, Pico Rivera, California
  - Research Site, San Diego, California
  - Research Site, Wildomar, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Maitland, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Smyrna, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Joliet, Illinois
  - Research Site, Greenwood, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, Farmington Hills, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington
  - Research Site, South Kirkland, Washington